CLINICAL TRIAL: NCT01754311
Title: Influence of IL28B Genetic Variation on the Phenotype Infection of HTLV-1
Acronym: HAMIL28B
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Laboratoire Cerba (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13/B/01
Record Dates: First submitted 2012-12-14; First posted 2012-12-21 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: HTLV-I Infections
Keywords: HTLV-I
MeSH Terms: conditions — HTLV-I Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HTLV-1 infected patients: HAM/TSP patients and HTLV-1 Asymtomatic patients
- control: Blood donors

SUMMARY:
Only 5 to 10% of patients infected with HTLV-1 develop a disease related to infection. The two most serious diseases are adult T-cell leukemia (ATL) and Tropical spastic paraparesis /HTLV-I-associated myelopathy (TSP / HAM). Factors influencing the development of TSP / HAM in the individual HTLV-1 are not yet completely understood. Patients TSP / HAM have a HTLV-1 proviral load (amount of virus) that is 6-10 times higher than seropositive asymptomatic.

Various studies have shown that the development of TSP / HAM in the subject HTLV-1 and its rapid evolution is partly attributed to the failure of the immune system that regulates viral replication and expression.

It has recently been shown that different versions of Single Nucleotide (human leukocyte antigen) rs12979860, located upstream of the gene for Interleukin 28B (IL28B), influenced the severity of infection with hepatitis C and effectiveness of treatment.

By analogy with hepatitis C, a Spanish (Treviño et al., 2012) examined this SNP(single nucleotide polymorphism) in 12 patients TSP / HAM and 29 asymptomatic HIV-positive. CT or TT genotype was statistically more frequent in the group TSP / HAM than in asymptomatic patients (80% versus 20%) and was associated with HTLV-1 proviral load higher.

We propose a broader group of patients in our population and Afro-Caribbean, to confirm the results of the latter study was conducted in a predominantly Latin American population.

ELIGIBILITY:
Inclusion Criteria :

HAM/TSP Patient:

* Age over 18 years
* Whose HAM/TSP was diagnosed on the criteria of Belem (De Castro-Costa et al., 2006)
* Follow regular consultation of Neurology of the University Hospital of Fort-de-France,
* Affiliate a system of social security (or entitled Beneficiary)
* Having agreed to participate in research by signing the consent form.

HTLV-1 asymptomatic patient:

* Age over 18 years
* Follow regular consultation of Neurology of the University Hospital of Fort-de-France,
* Do not show clinical signs of neurological impairment (a pyramidal syndrome with functional impairment clinic, genito-sphincter, motor deficits suggestive of polymyositis belts)
* Affiliate a system of social security (or entitled Beneficiary)
* Having agreed to participate in research by signing the consent form.

Blood donors:

* Respecting the eligibility criteria for blood donation
* Affiliated with the social security system (or entitled Beneficiary)
* Having agreed to participate in research by signing the consent form
* Serology HTLV-1 negative at the time of blood donation

Exclusion Criteria :

HAM/TSP Patient:

* Featuring an intricate polypathology may cast doubt on the responsibility of HTLV-1 in neurological symptoms,
* Infected with HIV or HBV or HCV
* Not affiliated to a social security (or entitled beneficiary)
* Do not sign the form for obtaining consent.

HTLV-1 asymptomatic patient:

* Infected with HIV or HBV or HCV
* Not affiliated to a social security (or entitled beneficiary)
* Do not sign the form obtaining informed consent.

Blood donors:

* Do not meet the eligibility criteria for blood donation
* Not affiliated to a social security (or entitled beneficiary)
* Do not sign the form obtaining informed consent
* Serology HTLV-1 positive or doubtful

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HTLV-1 infected patients :
  Adult, followed in consultation of Neurology of the University Hospital of Fort-de-France for their HTLV-1 infection.
  Blood Donors ; Adult, age 18 to 70 years coming to give their blood in one of building or mobile collection facilities of Martinique French Blood Establishement
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-06-24 (Actual)

PRIMARY OUTCOMES:
Presence of CT or TT allele for each participant | 30 days
  The participants will be followed until the end of the study ( with an expected average of 30 days after the inclusion).
  Explenations : each participant will have a blood sample who will be performed at the recruitement day (for génetics analysis) . After this first visit (recuitement visit) , each participant will have to perform an appointement with the ophtalmologic département ( recuperate datas about the presence or not of an uveitis and a keratoconjunctivitis)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Olindo, MD, Principal Investigator — University Hospital of Fort de France
Locations (2):
- Martinique (2):
  - University Hospital of Fort de France, Fort-de-France
  - French Blood Establishement, Fort-de-France